CLINICAL TRIAL: NCT03790826
Title: Chronic Indwelling Foley and Catheter Associated Trauma (CIF-CAT) Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nellie Medical, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CIFCAT-001
Record Dates: First submitted 2018-12-27; First posted 2019-01-02 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Bladder Infections and Inflammations
Keywords: bladder mucosal trauma
MeSH Terms: conditions — Cystitis; Inflammation | interventions — Cystoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cystoscopic Inspection (Experimental): Comparison of bladder damage with traditional Foley catheter and the Kohli Atraumatic catheter.
  Interventions: cystoscopy
  Interventions: Device: cystoscopy

INTERVENTIONS:
Device: cystoscopy — Comparison of bladder mucosa via cystoscopy.

SUMMARY:
To determine whether an indwelling low profile Kohli Atraumatic Catheter causes less macro-morphologic inflammation and edema to the bladder mucosa than a traditional indwelling Foley catheter as assess by computerized image analysis.

DETAILED DESCRIPTION:
The Kohli Atraumatic Catheter similarly aims to reduce bladder mucosal trauma with its low profile pancake shaped balloon versus the ovoid balloon of a traditional Foley catheter. The Kohli Atraumatic Catheter has a short, opened-ended tip that minimally protrudes through a patented low-profile donut-shaped balloon. The combination of the low profile and reduced tip length prevents the catheter from contacting the bladder walls and thereby minimize disruption of the bladder surface mucus layer and trauma to the urothelium - theoretically reducing the chance of bacterial invasion. A trial in which sheep were randomized to a traditional indwelling Foley catheter or a prototype Kohli Atraumatic Catheter demonstrated a dramatic reduction in both bladder wall trauma and edema. The ulcerated area dropped from 7.2% to 1.8% (75%) and the edema from 26.9% to 13.0% (52%).

Statistical Analysis To compare the effects of 2 catheter types, data will be analyzed using the general linear models tools from SAS/STAT software and presented as means ± standard error of the mean. The model will include 2 catheter types, inflamed vs non-inflamed areas, and their interactions.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women older than age 18
* Indwelling Foley urinary catheter for at least 30 days prior to entry with anticipation for continued indwelling urinary catheterization for at least 30 days after entry into the study.

Exclusion Criteria:

* Inability to provide informed consent
* Unwilling or medically inappropriate for cystoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Bladder mucosa damage assessment via computerized image analysis | 30 days
  Macro-morphologic inflammation and edema assessment of bladder mucosa using computerized image analysis.
  Image Analysis Technique Image of each bladder will be analyzed using FLIR Research IR Software (FLIR Systems Inc., Wilsonville, OR) to determine the proportion of inflamed areas characterized by red surface including hemorrhage and ulceration, and edema (eg, swollen smooth surface) out of total bladder area.

SECONDARY OUTCOMES:
Bladder mucosa damage urologist visual assessment | 30 days
  Visual macro-morphologic inflammation and edema assessment of bladder mucosa by experienced urologists familiar with the assessment of bladder diseases. Images and videos from a first visit where the traditional Foley catheter has been in place will be compared to those from a subsequent cystoscopy. Urologists will be blinded as to the catheter associated with each block of images captured during the cystoscopy.
Patient discomfort via Numeric Pain Rating Scale | 30 days
  A numeric pain rating scale chart will be completed by each patient for comparison of patient discomfort with a traditional indwelling Foley catheter in patients with chronic indwelling Foley catheters. The scale runs from 0 "No Pain" to 5 "Moderate Pain" and 10 "Worst Possible Pain." More information on the scale can be seen here "https://www.physio-pedia.com/Numeric_Pain_Rating_Scale" There are no Subscales and the marked score for first assessment will be compared to 2nd assessment to assess any changes in patient comfort with the two different catheters.

IPD SHARING:
Plan to Share IPD: No